CLINICAL TRIAL: NCT05188859
Title: Study of Sintilimab Combined With Anlotinib and Platinum-Containing Dual-Agent Chemotherapy as First Line Therapy in Malignant Pleural Mesothelioma: A Single Arm, Open-label, Prospective Phase II Trial
Brief Title: First Line Sintilimab Combined With Anlotinib and Platinum Doublet Chemotherapy in Malignant Pleural Mesothelioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jie Wang, Chief of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2950
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Mesothelioma, Malignant; Mesothelioma, Malignant Pleural; Mesothelioma Malignant Advanced
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Regimen:
  1. Sintilimab, 200mg, ivgtt d1, q3w, on a 21-day cycle, for a maximum of 24 months;
  2. Anlotinib, 12mg, po, qd, d1-14, q3w, on a 21-day cycle, for a maximum of 24 months;
  3. Pemetrexed, 500mg/m², ivgtt , d1, q3w, on a 21-day cycle;
  4. Cisplatin, 75mg/m2 , ivgtt, d1, q3w/Carboplatin, AUC 5.0, ivgtt, d1, q3w, on a 21-day cycle, 4-6 cycles.
  Interventions: Drug: Sintilimab+Anlotinib+Pemetrexed+Cisplatin

INTERVENTIONS:
Drug: Sintilimab+Anlotinib+Pemetrexed+Cisplatin — Sintilimab 200mg+Anlotinib 12mg+Pemetrexed 500mg/m²+Cisplatin 75mg/m2
  Other Names: S+A+PC

SUMMARY:
This study is a single-arm, open-lable, single-center phase II clinical trial for patients with advanced or metastatic pleural mesothelioma. The aim of this study was to observe and evaluate the efficacy and safety of Sintilimab combined with Anlotinib hydrochloride and platinum-containing dual-agent chemotherapy as first-line therapy in malignant pleural mesothelioma.

DETAILED DESCRIPTION:
Patients with advanced or metastatic (stage IIIB or IV) pleural mesothelioma who had not received previous systemic therapy were screened for eligible subjects to be eligible for enrollment after signing an written informed consent to receive Sintilimab combined with Anlotinib hydrochloride and platinum-containing dual-agent chemotherapy until disease progression (PD), intolerable toxicity, withdrawal of informed consent, initiation of other antineoplastic therapy, death or other situations for which protocol specified treatment should be discontinued (whichever occurs first). The maximum duration of treatment with Sintilimab is 24 months (in general).

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent before implementing any trial-related procedures;
* Age ≥ 18 years old.
* Histologically confirmed, unresectable or inoperable or locally advanced (IIIB stage), recurrent or metastatic (IV stage) malignant pleural mesothelioma.
* According to the modified version of the evaluation criteria for the efficacy of solid tumor (mRECIST1.1 ), patients have at least one imaging lesion can be measured;
* Patients have not received any systemic anti-tumor therapy for advanced/metastatic diseases in the past. Patients who have previously received platinum-containing adjuvant / neoadjuvant chemotherapy, or radical radiotherapy and chemotherapy for advanced diseases, such as the interval between disease progression or recurrence and the end of the last chemotherapeutic drug treatment at least 6 months, are allowed to be enrolled in this study.
* Patients with brain metastasis who are asymptomatic or stable after local treatment are allowed to be included in this study, as long as they meet the following conditions:

  1. There are measurable lesions outside the central nervous system.
  2. No central nervous system symptoms or no aggravation within at least 2 weeks.
  3. Those who do not need glucocorticoid therapy or stop glucocorticoid therapy within 7 days before the first study drug administration.
* Patients are allowed to receive palliative radiotherapy, but the end of radiotherapy is within 7 days before the administration of the first study drug.
* ECOG score 0-1 points;
* The expected survival time was > 3 months,
* For adequate organ function, the patients need to meet the following laboratory indexes:

  1. the absolute value of neutrophils (ANC) ≥ 1.5x109/L without granulocyte colony stimulating factor in the past 14 days.
  2. in the last 14 days without blood transfusion, the platelet count was ≥ 100x109/L.
  3. in the absence of blood transfusion or the use of erythropoietin in the past 14 days, hemoglobin > 9g/dL;
  4. Total bilirubin ≤ 1.5 × normal upper limit (ULN); for example,if total bilirubin > 1.5 × ULN but direct bilirubin ≤ ULN is also allowed to enter the group
  5. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (patients with liver metastasis allow ALT or AST ≤ 5 × ULN).
  6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥ 60ml;
  7. Coagulation function is good, defined as international standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
  8. Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is beyond the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled.
  9. Myocardial enzyme spectrum is within the normal range (if the researchers comprehensively judge that there is no clinical significance of simple laboratory abnormalities can also be included in the group); (optional)
* For female patients at childbearing age, they should undergo a urine or serum pregnancy test within 3 days before receiving the first study drug administration (day 1 of cycle 1) and the results be negative. If the urine pregnancy test results cannot be confirmed as negative, a blood pregnancy test is required. Women of non-childbearing age are defined as at least 1 year after menopause or have undergone surgical sterilization or hysterectomy.
* If there is a risk of pregnancy, all patient (male or female) are required to use contraception with an annual failure rate of less than 1% during the entire treatment period until 120 days after the last study drug administration (or 180 days after the last chemotherapy drug administration).

Exclusion Criteria:

* Diagnosis of malignant diseases other than malignant pleural mesothelioma (excluding radical skin basal cell carcinoma, skin squamous cell carcinoma, and / or radical resection of carcinoma in situ) within 5 years before the first administration
* Currently participating in interventional clinical research treatment, or receiving other research drugs or using research instruments within 4 weeks before the first administration;
* Previous usage of the following treatments: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs, for another stimulating or synergistic inhibition of T cell receptors (for example, CTLA-4, OX-40, CD137) drug;
* Within 2 weeks before the first administration, they received systemic systemic therapy with anti-tumor indications of proprietary Chinese medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, except for controlling local use of pleural effusion)
* Active autoimmune diseases requiring systemic treatment (such as the use of disease-relieving drugs, glucocorticoids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapy (such as thyroxine, insulin or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy.
* The patients are received systemic glucocorticoid therapy (excluding nasal, inhaled or other topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first administration.

Note: The use of physiological doses of glucocorticoids (≤10 mg/day prednisone or equivalent drugs) is allowed;

* There are clinically uncontrollable pleural effusion / ascites (patients who do not need drainage or stop drainage for 3 days without a significant increase in effusion can be enrolled in the group)
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Those who are known to be allergic to the active ingredients or excipients of Sintilimab in this study.
* Patients with multiple factors affecting oral drugs (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.)
* Symptomatic or uncontrolled brain metastasis;
* Active hemoptysis (at least 2.5ml or 1/2 teaspoon of blood was spit out at a time) 3 months before the first study drug administration;
* Imaging showed that there were tumors invading / infiltrating large blood vessels or bleeding tendency assessed by researchers or radiologists;
* Received major surgery (except for surgery for the purpose of biopsy) within 4 weeks before the first study drug administration, or is expected to undergo major surgery during the study period;
* Severe unhealed wound ulcers or fractures;
* Minor surgery was performed within 48 hours before first receiving the study drug (outpatient / inpatient surgery requiring local anesthesia, including central venous catheterization);
* Use aspirin (>325 mg/day) or other non-steroidal anti-inflammatory drugs that are known to inhibit platelet function for 10 consecutive days (within 10 days before receiving the first dose of study drug) at present or in the near future;
* Current or recent treatment with full-dose oral or parenteral anticoagulants or thrombolytic agents for 10 consecutive days (within 10 days before receiving the first study drug) Note: Prophylactic use of low-dose anticoagulants is permitted: low-dose warfarin (≤ 1mg/d) is allowed for preventive purposes on the premise that the international standardized ratio of prothrombin time (INR) ≤ 1.5. Low-dose heparin (≤ 12000 U/e d) or low-dose aspirin (≤ 100mg/d).
* Hereditary bleeding tendency or coagulation dysfunction, or history of thrombosis;
* Did not fully recover from toxicity and / or complications caused by any intervention (i.e., ≤ level 1 or reached baseline, excluding fatigue or hair loss) before starting treatment;
* Known human immunodeficiency virus (HIV) infection history (i.e. HIV 1/2 antibody positive)
* Untreated active hepatitis B (defined as HBsAg positive and the number of HBV-DNA copies detected is greater than the upper limit of the normal value of the laboratory in the research center).

Note: hepatitis B subjects who meet the following criteria can also be enrolled in the group:

1. Before the first administration, the HBV viral load is less than 1000 copies/ml (200 IU/ml), and the patients should receive anti-HBV treatment during the entire study drug treatment period to avoid viral reactivation;
2. For patients with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), there is no need to receive preventive anti-HBV therapy. However, the virus needs to be closely monitored for reactivation

   * Active HCV infection subjects (HCV antibody positive and HCV-RNA level higher than the lower limit of detection)
   * Live vaccine is given within 30 days before the first administration (cycle 1, day 1).

Note: It is allowed to receive inactivated virus vaccine for seasonal influenza within 30 days before the first administration; however, it is not allowed to receive live attenuated influenza vaccine for intranasal administration..

* Pregnant or lactating women;
* There are any serious or uncontrollable systemic diseases, such as

  1. significant abnormalities in rhythm, conduction, or morphology of resting electrocardiogram and serious and uncontrollable symptoms, such as complete left bundle branch block, second-degree cardiac block, ventricular arrhythmia or atrial fibrillation.
  2. unstable angina pectoris, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) grade ≥ 2;
  3. any arterial thrombosis, embolism or ischemia occurred within 6 months before treatment, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack;
  4. Blood pressure control is not satisfactory (systolic blood pressure > 140mmHg, diastolic blood pressure > 90mmHg).
  5. within 1 year before the first administration, there is a history of non-infectious pneumonia requiring glucocorticoid treatment, or currently there is clinically active interstitial lung disease;
  6. active pulmonary tuberculosis;
  7. active or uncontrolled infections requiring systemic treatment;
  8. clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction.
  9. liver diseases such as liver cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L);
  11. patients with urinary protein ≥ + + and confirmed 24-hour urinary protein quantity > 1.0g;
  12. patients with mental disorders and unable to cooperate with treatment
* At the discretion of the investigator, there are patients with serious concomitant disease that compromises patient safety or affects the patient's completion of the study; The investigator believes that there are other potential risks and is not suitable for participation this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months after the final enrollment
  Objective Response Rate（ORR）according to mRECIST 1.1 standard

SECONDARY OUTCOMES:
DOR | 24 months
  Duration of remission
DCR | 24 months
  Disease Control Rate
PFS | 24 months
  Progression Free Survival
OS | 24 months
  Overall Survival
AE | 24 months
  Adverse event
SAE | 24 months
  Incidence and Severity of Serious Adverse Event
Lab indicators | 24 months
  Abnormal values of laboratory indicators

CONTACTS AND LOCATIONS:
Overall Officials: Wang, MD,PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Shanxi Provincial Cancer Hospital/ Shanxi Hospital Affiliated to Cancer Hospital, Chinese Academy of Medical Sciences/Cancer Hospital Affiliated to Shanxi Medical University, Taiyuan, Shanxi
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No